CLINICAL TRIAL: NCT01406522
Title: Tacrine Effects on Cocaine Self-Administration and Pharmacokinetics
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: One of the study medications, tacrine, is no longer clinically available
Sponsor: Midwest Biomedical Research Foundation (Other)
Responsible Party: Principal Investigator, KENNETH GRASING, Director, Substance Abuse Research Laboratory, Midwest Biomedical Research Foundation
Organization: Midwest Veterans' Biomedical Research Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21DA029787 (NIH)
Record Dates: First submitted 2011-07-28; First posted 2011-08-01 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Cocaine Dependence
Keywords: Acetylcholine; Cholinesterases; Cocaine; Self-Administration
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Tacrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral placebo (Placebo Comparator): Inactive treatment
  Interventions: Drug: Oral placebo
- Oral tacrine (Experimental): Oral tacrine
  Interventions: Drug: Oral tacrine

INTERVENTIONS:
Drug: Oral tacrine — Tacrine, 160 mg per day, four times daily
  Arms: Oral tacrine
Drug: Oral placebo — Microcrystalline cellulose
  Arms: Oral placebo

SUMMARY:
No medications are currently available for treatment of psychostimulant addiction, a compulsive preoccupation with use of cocaine and related compounds. Tacrine, a medication that is currently prescribed for Alzheimer's disease, can decrease the amount of cocaine injections that laboratory animals choose to inject by vein. This project will determine if tacrine can also decrease cocaine-motivated behavior for human subjects in a laboratory setting.

DETAILED DESCRIPTION:
Background Reinforcing effects of cocaine are believed to arise through release of dopamine (DA) at the nucleus accumbens by neurons in the ventral tegmental area. Activation of cholinergic receptors on the cell bodies of these neurons can enhance DA release. Elevated levels of acetylcholine (ACh) in the nucleus accumbens may also serve to inhibit appetitive behaviors. Cholinesterase inhibitors such as tacrine increase synaptic levels of ACh by preventing its inactivation by acetylcholinesterase (AChE) or butyrylcholinesterase (BuChE), and can improve learning and memory. In animals, cholinesterase inhibitors can attenuate cocaine self-administration and conditioned place preference. Tacrine is a centrally acting, reversible inhibitor of AChE and BuChE that is approved for treatment of Alzheimer's disease. In addition to its effects on the cholinergic system, tacrine can potentiate the actions of monoamines, including DA. Although use of tacrine has declined because of requirements for monitoring of potential liver toxicity and pharmacokinetics that necessitate multiple daily doses, it is more potent than other cholinesterase inhibitors in attenuating cocaine self-administration in animals. Pretreatment with tacrine can produce long-lasting reductions in cocaine-reinforced behavior in rats, described as persistent attenuation (cocaine self-administration is decreased by more than 80% over a period of three days during which no additional cholinesterase inhibitor is administered, see Figure 1). No previous studies have evaluated whether tacrine can modify the effects of cocaine in humans.

Rationale To our knowledge, tacrine is the only compound that can produce persistent attenuation in rats treated with clinically relevant doses. If similar effects were observed in humans, this would lead to an important paradigm shift for substance abuse treatment, in that large reductions in cocaine-reinforced behavior could be produced without the need for continuous dosing with a medication. This scenario could remove the requirement for continued compliance with oral dosing in some patients with its associated potential for toxicity.

Specific Aims:

1. Evaluate whether tacrine treatment causes persistent attenuation of cocaine-reinforced behavior in humans.
2. Determine the effectiveness of pretreatment with tacrine in attenuating cocaine-induced craving.
3. Evaluate plasma levels of cocaine and characterize the bioavailability of tacrine in individual patients.

Methods This is a randomized, double-blind, double-dummy, placebo-controlled, inpatient, single-center, parallel-group evaluation of the potential for oral tacrine to modify cocaine self-administration, cocaine-induced craving, and the pharmacokinetics of cocaine and tacrine. To evaluate the occurrence of persistent attenuation, the subjective and reinforcing effects of intravenous cocaine will be determined during oral treatment and three days following its discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV-TR criteria for cocaine abuse or dependence, with at least one cocaine-positive urine specimen within the six weeks prior to enrollment.
* Has used cocaine for a duration of at least 6 months, with at least weekly use during the last 30 days by a rapid route of administration (either smoked or intravenous injection).
* Is male or female, between 21 and 50 years old.

Exclusion Criteria:

* Has a history of a medical adverse reaction to cocaine or other psychostimulants, including loss of consciousness, chest pain, cardiac ischemia, or seizure.
* Has any current Axis I psychiatric disorder other than drug abuse or dependence.
* Meets DSM-IV-TR criteria for dependence on opiates, benzodiazepines, alcohol, or other sedative-hypnotics.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2013-09 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Decreased cocaine-reinforced behavior | Day 9 of treatment
  participants will make a series of choices between vouchers with an ascending monetary value and intravenous injections of cocaine

SECONDARY OUTCOMES:
Changes in cocaine pharmacokinetics | Day 9 of treatment
  Plasma levels of cocaine and metabolites will be determined by liquid chromatography-tandem mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth W Grasing, M.D., Principal Investigator — Kansas City VA Medical Center
Locations (1):
- Kansas City VA Medical Center, Kansas City, Missouri, United States

REFERENCES:
- [Background] Grasing K, He S, Yang Y. Dose-related effects of the acetylcholinesterase inhibitor tacrine on cocaine and food self-administration in rats. Psychopharmacology (Berl). 2008 Jan;196(1):133-42. doi: 10.1007/s00213-007-0944-3. Epub 2007 Oct 5. PMID 17917719
- [Background] Grasing K, He S, Yang Y. Long-lasting decreases in cocaine-reinforced behavior following treatment with the cholinesterase inhibitor tacrine in rats selectively bred for drug self-administration. Pharmacol Biochem Behav. 2009 Nov;94(1):169-78. doi: 10.1016/j.pbb.2009.08.004. Epub 2009 Aug 19. PMID 19698738